CLINICAL TRIAL: NCT03624114
Title: Prediction of Sphenoid Septation in Magnetic Resonance Imaging Compared With Computed Tomography and Intraoperative Findings During Endoscopic Pituitary Adenoma Surgery - a Prospective Observational Study
Brief Title: Prediction of Sphenoid Septation in MRI Compared With CT and Intraoperative Findings During Endoscopic Pituitary Adenoma Surgery
Acronym: Scope
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-00065; ch18Roethlisberger
Record Dates: First submitted 2018-08-07; First posted 2018-08-09 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Pituitary Adenoma
Keywords: pituitary adenoma surgery; endoscopic transsphenoidal surgery; sphenoid septation
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: comparison of data from MRI with data from CT compared with intraoperative data from endoscopic pituitary adenoma surgery — A comparison of MRI with CT of the skull base or paranasal sinuses and intraoperative Video documentation of the anatomical site will be used.

SUMMARY:
To investigate whether MRI is able to predict the exact anatomy and topography of the sphenoid sinus and its relationship to the sellar, parasellar und paraclinoid region and where CT yields more detailed information for the surgeon before trans-sphenoidal pituitary adenoma surgery.

DETAILED DESCRIPTION:
The current research project addresses the question whether MRI alone is sufficient for preoperative planning and computer-assisted surgery (CAS) during standard trans-sphenoidal pituitary surgery and if situations can be identified, where additional CT yields more information for the surgeon.

A comparison of MRI with CT of the skull base or paranasal sinuses and intraoperative Video documentation of the anatomical site will be used.

50 patients operated the University hospital of Basel [USB] (Centre A) are consecutively included into the prospective part of the study. MRI is used to assess the standardized variables, confirmed by CT. Additionally, for the 50 prospectively collected patients, neuroimaging results are correlated with intraoperative evaluation during endoscopic trans-sphenoidal surgery or post-hoc with video analysis of the performed surgery.

Between 20-50 patients operated at the University of Malaya Medical Centre [UMMC] and Specialist Centre [UMSC] (Centre B)will be included retro- and prospectively . MRI is used to assess the standardized variables and the results are correlated with intraoperative evaluation during endoscopic trans-sphenoidal surgery or post-hoc with video analysis of the performed surgery.

ELIGIBILITY:
Inclusion Criteria:

* lndicated trans-nasal trans-sphenoidal surgery for an anterior skull base tumour with preoperative baseline MRI (Centre A and B) and baseline CT (Centre A).

Exclusion Criteria:

* Previous trans-sphenoidal surgery
* Patients without CT, MRI or intraoperative endoscopic video

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with sphenoidal surgery for an anterior skull base tumor with preoperative MRI, CT and intraoperative video during endoscopy (Centre A) and preoperative MRI and intraoperative video during endoscopy (Centre B).
  Consecutive recruitment of patients with planned endonasal endoscopic anterior skullbase tumors in daily clinical practice in both centres (A and B).
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Posterior Insertion Site of the sphenoid septum at Cavernous Carotid and/or Optico-Carotid-Recess | duration of endoscopic transsphenoidal surgery
  To compare the relative performance of the MRI and the CT scan regarding posterior insertion site of the sphenoid septum at cavernous carotid and/or optico-carotid-recess. Neuroimaging results are correlated with intraoperative evaluation during endoscopic transsphenoidal surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Röthlisberger, Dr. med, Principal Investigator — University Hospital, Basel, Switzerland
Locations (2):
- University of Malaya Medical Center and Specialist Center, Petaling Jaya, Malaysia
- University Hospital Basel, Neurochirurgie und Spinale Chirurgie, Basel, Switzerland